CLINICAL TRIAL: NCT01337570
Title: A Multi-Centre, Randomised, Double-Blind, Placebo-Controlled Phase III Safety and Efficacy Trial of a Vaginal Matrix Ring With Dapivirine for the Prevention of HIV-1 Infection in Women
Brief Title: A Safety and Efficacy Trial of Dapivirine Vaginal Ring in Africa
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Sponsor: International Partnership for Microbicides, Inc. (Industry)
Responsible Party: Annalene Nel, MBChB, PhD, International Partnership for Microbicides, Inc.
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: IPM 009A
Record Dates: First submitted 2011-04-13; First posted 2011-04-19 (Estimated); Last update posted 2012-06-11 (Estimated); Status verified 2012-06

CONDITIONS: HIV Infections
Keywords: HIV Infections; Anti-HIV agents; HIV-1
MeSH Terms: conditions — HIV Infections | interventions — Dapivirine

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Dapivirine (Experimental): Vaginal ring containing 25mg of dapivirine
  Interventions: Other: Dapivirine; Drug: Dapivirine
- Placebo Ring (Placebo Comparator): Vaginal ring containing no drug substance
  Interventions: Other: Placebo

INTERVENTIONS:
Other: Dapivirine — Vaginal ring containing 25mg dapivirine; one ring inserted every 28 days for at least 15 months
  Arms: Dapivirine
Other: Placebo — Vaginal Ring containing no drug substance
  Arms: Placebo Ring
Drug: Dapivirine
  Arms: Dapivirine

SUMMARY:
This is a double-blind, randomized, placebo-controlled Phase III study to assess the safety and efficacy of a silicone elastomer vaginal ring containing 25mg of dapivirine.

ELIGIBILITY:
Inclusion Criteria:

* Women >18 and <40 years of age who can provide informed consent
* Available for all visits and consent to follow all procedures scheduled for the trial
* Generally healthy and self-reported sexually active (defined as an average of at least one penetrative penile vaginal coital act per month for the last 3 months prior to enrolment)
* HIV-negative as determined by the HIV algorithm applied at screening and enrolment
* On a stable form of contraception as defined within section 5.4 and willing to continue on stable contraception for the duration of the clinical trial;
* Asymptomatic for genital infections at the time of enrolment (if a woman is diagnosed with any clinically significant treatable STI, she must have initiated treatment at least 1 week prior to enrolment and have completed the full course of treatment)
* Willing to answer questions about adherence, sexual behaviour, vaginal practices and ring acceptability;
* Willing to provide adequate locator information for trial retention purposes and be reachable per local standard procedures (e.g., by home visit or telephone; or via family or close neighbour contacts [confidentiality to be maintained])
* Willing to refrain from participation in another research trial using drugs, vaccines, medical devices, microbicides or oral pre-exposure prophylaxis investigational drugs for the duration of the IPM 009A trial;
* In the absence of the use of exogenous hormone(s), have a self-reported regular menstrual cycle defined as having a minimum of 21 days and a maximum of 35 days between menses;
* Willing to refrain from use of vaginal products or objects including spermicides, tampons, female condoms, cotton wool, rags, diaphragms, cervical caps (or any other vaginal barrier method), douches and drying agents within 14 days from enrolment and for the duration of the trial.

Exclusion Criteria:

* Currently pregnant or last pregnancy within 3 months prior to screening;
* Currently breast-feeding
* Participated in another research trial using drugs, medical devices, microbicides or oral pre-exposure prophylaxis agents within 60 days prior to screening
* Previously participated or currently participating in any HIV vaccine trial
* Untreated, clinically significant urogenital infections (either symptomatic or asymptomatic), e.g., urinary tract or other sexually transmitted infections, or other gynaecological symptoms within 1 week prior to enrolment
* History of significant urogenital or uterine prolapse, undiagnosed vaginal bleeding, urethral obstruction, incontinence or urge incontinence
* Any gynaecological surgery within 90 days prior to enrolment
* Any Grade 3 or 4 baseline haematology, chemistry or urinalysis laboratory value according to the DAIDS Table for Grading Adverse Experiences, or clinically significant Grade 2 findings
* Any history of anaphylaxis or severe allergy resulting in angioedema; or a history of sensitivity/allergy to latex or a silicone elastomer
* Any history of diabetes mellitus and chronic use of oral steroid therapy and any uncontrolled serious chronic or progressive disease
* Cervical cytology at screening that requires cryotherapy, biopsy, treatment (other than for infection), or further evaluation [this includes any findings of atypical squamous cells of undetermined significance (ASCUS)]
* Any condition(s) that, in the opinion of the investigator, might put the participant at risk, or interfere with the trial objectives, or adherence to trial requirements

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2011-07; Primary Completion 2014-07 (Estimated); Study Completion 2014-07 (Estimated)

PRIMARY OUTCOMES:
Efficacy as determined by the proportion of women in each arm HIV-1 seroconversion rate per person-years of product use, measured at the end of the investigational product use period. | 15 months
  The primary endpoint is HIV-1 seroconversion measured by rapid and specialized laboratory tests according to a comprehensive HIV testing algorithm. This algorithm employs a series of high specificity and high sensitivity immunoassay-based HIV blood tests that minimize the chance of false positive results to determine if a subject is positive for HIV. Endpoint confirmation of HIV infection is by Western blot.
Safety as determined by grade 3 and 4 AE's, clinically significant grade 2 laboratory findings (based on DAIDS grading) and all serious AE's. | 15 months
  This will be measured by self-reports, physical examination, safety laboratory tests and other specialised investigations.

SECONDARY OUTCOMES:
Adherence to the protocol-specific product regimen as determined by self-reported diary cards and questionnaires. | 15 months
The incidence of curable STI's or pregnancy as determined by STI testing and pregnancy testing. | 15 months

CONTACTS AND LOCATIONS:
Overall Officials: Annalene Nel, Study Director — Beijing Immupeutics Medicine Technology Limited
Locations (5):
- College of Medicine - Johns Hopkins Project (JHP), Blantyre, Malawi
- African University Clinical Research Centre, Kigali, Rwanda
- South Africa (2):
  - Qhakaza Mbokodo, Ladysmith, KwaZulu-Natal
  - Madibeng Centre for Research (MCR), Brits
- African University Clinical Research Centre, Mutare, Zimbabwe